CLINICAL TRIAL: NCT04855019
Title: Comparison of Combined Suprascapular and Axillary Nerve Blocks With Periarticular Injection for Analgesia in Arthroscopic Shoulder Surgery
Brief Title: Post Surgical Pain in Arthroscopic Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Ayhan ŞAHİN, Principal Investigator, Namik Kemal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Shoulder Surgery
Record Dates: First submitted 2021-04-17; First posted 2021-04-22 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-11

CONDITIONS: Total Shoulder Arthroplasty
Keywords: shoulder arthroplasty; suprascapular block; axillary nerve block; periarticular injection; ultrasound

STUDY DESIGN:
Intervention Model Description: prospective randomized trial, To compare the suprasacuplar-axillary nerve block combined with the periarticular injection method in shoulder arthroscopy cases.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- periarticular injection group (PI) (Active Comparator): the group to be given a periarticular injection by an orthopedist
  Interventions: Procedure: shoulder periarticular injection, suprascapular and axillary nerve block
- Combined suprascapular-axillary nerve block group (CSAB) (Active Comparator): the group in which an anesthesiologist will perform combined suprascapular axillar border block under ultrasound guidance
  Interventions: Procedure: shoulder periarticular injection, suprascapular and axillary nerve block

INTERVENTIONS:
Procedure: shoulder periarticular injection, suprascapular and axillary nerve block — In the PI group, a mixture of 30 ml bupivacaine 0.5% and 30 ml saline solution will be injected by the orthopedist after the wound is closed.
  In the CSAB group, a total of 20 ml 0.5% bupivacaine, 10 ml to the suprascapular notch, 10 ml to the axillary nerve, will be administered preoperatively by the anesthesiologist under ultrasound guidance.

SUMMARY:
Postoperative multimodal analgesia methods occupy an essential place in modern anesthesia. The postoperative results of opioid analgesia are now at the bottom of the current problems due to its side effects. Longer-acting local anesthetics are now effective agents of analgesia.

Investigators aimed to compare the two routine methods. Ultrasonic nerve blocks are the most important of multimodal analgesia in modern anesthesia. Suprascapular and axillary nerve blocks are routinely used as a safe method. It is a routine method used by periarticular local anesthetic surgeons.

İnvestigators decided to compare which method effectively follows these two methods with the postoperative 24 pain scale method.

DETAILED DESCRIPTION:
This randomized trial aims to assess if a combined suprascapular-axillary nerve block (CSAB) to periarticular injection (PI) treated pain after arthroscopic shoulder surgery. Secondary endpoints included opioid consumption, discomfort associated with muscle weakness, and patient satisfaction.

sixty patients undergoing arthroscopic shoulder surgery will be randomized to receive ultrasound-guided CSAB (n = 30) or PI (n = 30). Pain intensity at rest and discomfort were recorded upon arrival in the recovery room, discharge to the ward, and at 4, 8, and 24 hours after surgery. Tramadol consumption was recorded for the first 24 hours. Patient satisfaction data will be recorded on the second postoperative day.

Using a computer-generated random allocation sequence (created by the study statistician), patients will randomly be assigned to ultrasound-guided SAB (n = 30) or PI(n = 30). Allocation numbers will be sealed in an opaque envelope opening in sequence by an independent anesthesiologist who will not assess outcomes. Outcome assessors will be blinded to treatment allocation.

After eligible patients are identified from the registry, patient charts were prospectively a blind orthopedist would collect data. Demographic data including sex, age, body mass index, surgical procedure, and complications will be recorded. Primary outcome measures were numeric rating scale pain scores and 24-hour postoperative opioid consumption. Pain scores will be recorded immediately before surgery, immediately following surgery in the postanesthesia recovery unit, and 24 hours postoperatively. Total opioid consumption will also be recorded for the first 24 hours following surgery. Secondary outcome measures included length of surgery, operating room time, perioperative anesthesia time, blood loss, hospital length of stay, and intraoperative and 30-day postoperative complication rates. Postoperative complications were further categorized as nerve-related, cardiopulmonary, and musculoskeletal (fracture or tendon rupture).

Statisticians will compare statistics between groups using a 2-sample t-test for normally distributed variables. The Wilcoxon rank-sum test will be used for non-normally distributed variables. A general linear model with correlated errors was used to account for repeated pain score assessments over time for each subject. The Fisher exact test will be used for categorical variables. Summary statistics will be reported as the mean and standard deviation for data analyzed using the 2-sample t-test and general linear models. The median and 25th and 75th percentiles will be reported for the Wilcoxon rank-sum test. The frequency (i.e., n) and percentage will be reported for data analyzed using the Fisher exact test. A P value of .05 will be designated as the threshold for statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Being in the age range of 18-65
* agree to participate in the study

Exclusion Criteria:

* diabetic patients
* chronic opioid use
* patients with sensitivity to local anesthetics
* patients with neuropathy
* Patients who cannot use the PCA
* cases returning to open surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Change from the baseline 11 point NRS (numeric rating Scala) Scala | 0 to 24 hours
  Possible scores range from 0 (no pain) to 10 ( worst possible pain). Change for 24 Hours.
Total opioid consumption, from the moment of exit from the operation to the 24th hour | 0 to 24 hours
  Each patient will be fitted with a patient controlled analgesia (PCA) device. The total tramadol requirement for both groups will be calculated.

SECONDARY OUTCOMES:
nausea and vomiting | 0 to 24 hours
  Data will be recorded in the postoperative period, in the form of present or not.

CONTACTS AND LOCATIONS:
Overall Officials: M.Cavidan ARAR, Study Chair — Prof.
Locations (1):
- Namık Kemal University, Tekirdağ, Süleymanpaşa, Turkey (Türkiye)